CLINICAL TRIAL: NCT00705874
Title: A Phase I Open Label, Multicenter, Dose-Escalation Study to Determine the Maximum Tolerated Dose, Dose Limiting Toxicity, Safety and Pharmacokinetics of CGC-11047 When Used in Individual Combinations With 1) Gemcitabine or 2) Docetaxel or 3) Bevacizumab or 4) Erlotinib or 5) Cisplatin or 6) 5-Flurouracil or 7) Sunitinib in Patients With Advanced Solid Tumors or Lymphoma
Brief Title: Study of CGC-11047 When Used in Individual Combinations With 1) Gemcitabine or 2) Docetaxel or 3) Bevacizumab or 4) Erlotinib or 5) Cisplatin or 6) 5-Flurouracil or 7) Sunitinib in Patients With Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Progen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 47-01-002
Record Dates: First submitted 2008-06-23; First posted 2008-06-26 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-06

CONDITIONS: Cancer
Keywords: cancer; advanced cancer; solid tumors; lymphoma; CGC-11047
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — CGC 11047; Gemcitabine; Docetaxel; Bevacizumab; Erlotinib Hydrochloride; Cisplatin; Leucovorin; Fluorouracil; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 (Experimental): CGC-11047 in combination with Gemcitabine
  Interventions: Drug: CGC-11047 and gemcitabine
- 2 (Experimental): CGC-11047 in combination with Docetaxel
  Interventions: Drug: CGC-11047 and docetaxel
- 3 (Experimental): CGC-11047 in combination with Bevacizumab
  Interventions: Drug: CGC-11047 and bevacizumab
- 4 (Experimental): CGC-11047 in combination with Erlotinib
  Interventions: Drug: CGC-11047 and erlotinib
- 5 (Experimental): Cisplatin: 80 mg/m2 administered IV over 1 hour once every 28 days. CGC-11047 will be administered on Days 1, 8 and 15 of a 28 day cycle.
  Interventions: Drug: CGC-11047 and cisplatin
- 6 (Experimental): CGC-11047 in combination with 5-Flurouracil / Leucovorin
  Interventions: Drug: CGC-11047 and 5-flurouracil / leucovorin
- 7 (Experimental): CGC-11047 in combination with Sunitinib
  Interventions: Drug: CGC-11047 and sunitinib

INTERVENTIONS:
Drug: CGC-11047 and gemcitabine — Gemcitabine: (Closed to enrollment) 1,000 mg/m2 administered IV over 30 minutes on Days 1, 8 and 15 of a 28-day cycle. CGC-11047 will only be given on days 1 and 15 of each cycle and will start at dose level -1 (50 mg).
  Other Names: Gemzar
  Arms: 1
Drug: CGC-11047 and docetaxel — Docetaxel: (Closed to enrollment) 75 mg/m2 administered IV over 60 minutes every 21 days. CGC-11047 will be administered only on Day 1 of each 21-day cycle and will start at dose level -1 (50 mg).
  Other Names: Taxotere
  Arms: 2
Drug: CGC-11047 and bevacizumab — Bevacizumab: 5 mg/kg administered IV once every 14 days. CGC-11047 will be administered on Days 1, 8 and 15 of a 28 day cycle.
  Other Names: Avastin
  Arms: 3
Drug: CGC-11047 and erlotinib — Erlotinib: 150 mg taken orally every day of each 28-day cycle. CGC-11047 will be administered on Days 1, 8 and 15 of a 28 day cycle.
  Other Names: Tarceva
  Arms: 4
Drug: CGC-11047 and cisplatin — Cisplatin: 80 mg/m2 administered IV over 1 hour once every 28 days. CGC-11047 will be administered on Days 1, 8 and 15 of a 28 day cycle.
  Arms: 5
Drug: CGC-11047 and 5-flurouracil / leucovorin — 5-Flurouracil / Leucovorin: Leucovorin 500 mg/m2 IV over 2 hours with 5 - FU 500 mg/m2 IV bolus starting 1 hour into leucovorin infusion weekly for 6 wks, repeated every 56 days. CGC-11047 will be administered on Days 1, 8 and 15 of a 28 day cycle.
  Other Names: 5-FU; Florouracil; Efudix
  Arms: 6
Drug: CGC-11047 and sunitinib — Sunitinib: 50 mg orally once daily, 4 weeks on treatment followed by 2 weeks off (42 day cycle). CGC-11047 will be administered on Days 1 and 8 of a 21 day cycle.
  Other Names: Sutent
  Arms: 7

SUMMARY:
This study will aims to determine the maximum tolerated dose of CGC-11047 when used in individual combinations with gemcitabine, or docetaxel, or bevacizumab, or erlotinib or cisplatin or 5-flurouracil or sunitinib in one of 7 treatment arms. The dose of CGC-11047 will be escalated until the maximum tolerated dose is established.

DETAILED DESCRIPTION:
This study will use a dose escalation design to determine the MTD of CGC-11047 when used in individual combinations with gemcitabine, or docetaxel, or bevacizumab, or erlotinib or cisplatin or 5-flurouracil or sunitinib in one of 7 treatment arms. The dose of CGC-11047 will be escalated in cohorts of 3 patients and dose escalation can proceed in each treatment group independent of dose escalation in the other treatment groups. CGC-11047 will be administered IV over 60 minutes and the doses of gemcitabine, docetaxel, bevacizumab, cisplatin, 5-flurouracil or sunitinib will remain fixed according to their respective product labeling.

ELIGIBILITY:
Inclusion Criteria:

* non-hematological advanced solid tumor malignancy or lymphoma where no curative therapy exists in which monotherapy with gemcitabine or docetaxel or bevacizumab or erlotinib or cisplatin, or 5-flurouracil or sunitinib would otherwise be warranted.
* measurable disease based on radiographic evaluation or elevated tumor markers.
* ECOG - 0 or 1 (KPS >70).
* Life expectancy > 3 months.

Exclusion Criteria:

* chemotherapy within 21 days or radiotherapy within 4 weeks prior to entering the study
* known active brain metastases or leptomeningeal carcinomatosis.
* history of a myocardial infarction within the prior 6 months or, hospitalizations for congestive heart failure within the prior 6 months, or active treatment for uncontrolled cardiac arrhythmias
* clinically significant gastrointestinal tract hemorrhage, requiring transfusion therapy, within the prior 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2006-05; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Stephenson, MD, Principal Investigator — Cancer Centres of the Carolinas, Greenville, SC 29605
Locations (12):
- United States (12):
  - Rocky Mountain Cancer Centre, Denver, Colorado
  - Cancer Centres of Florida, Ocoee, Florida
  - Central Indiana Cancer Centres, Indianapolis, Indiana
  - Comprehensive Cancer Centres of Nevada, Las Vegas, Nevada
  - New York Oncology Hematology PC, Albany, New York
  - Dayton Oncology and Hematology, PA, Kettering, Ohio
  - Cancer Centres of the Carolinas, Greenville, South Carolina
  - Texas Oncology, PA, Dallas, Texas
  - Tyler Cancer Centre, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer Specialists - Vancouver Cancer Centre, Vancouver, Washington
  - North Star Lodge Cancer Centre, Yakima, Washington

REFERENCES:
- See also: Progen Pharmaceuticals website — http://www.progen.com.au

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was June 2006 through March 2011, with last patient being treated May 2011. Patients were recruited through oncology clinics.
Pre-assignment Details: There was no run-in phase. Patients were assigned to treatment arm based on their cancer type and which standard of care therapy was appropriate based on Investigators' discreation.
Groups:
- PG11047/Gemcitabine: PG-11047 (infusion on Days 1 and 15 of each cycle) in combination with Gemcitabine (1,000 mg/m2 administered IV over 30 minutes on Days 1, 8 and 15 of a 28-day cycle).
- PG11047/Docetaxel: PG-11047 (infusion on Day 1 of each 21 day cycle) in combination with Docetaxel (75 mg/m2 administered IV over 60 minutes every 21 days).
- PG11047/Bevacizumab: PG-11047 (infusion on Days 1, 8 and 15 of a 28 day cycle) in combination with Bevacizumab (5 mg/kg administered IV once every 14 days).
- PG11047/Erlotinib: PG-11047 (infusion on Days 1, 8 and 15 of a 28 day cycle) in combination with Erlotinib (150 mg taken orally every day of each 28-day cycle).
- PG11047/Cisplatin: Cisplatin: 80 mg/m2 administered IV over 1 hour once every 28 days. PG-11047 will be administered by infusion on Days 1, 8 and 15 of a 28 day cycle.
- PG11047/5-Flurouracil: PG-11047 (infusion on Days 1, 8 and 15 of a 28 day cycle) in combination with 5-Flurouracil / Leucovorin (Leucovorin 500 mg/m2 IV over 2 hours with 5 - FU 500 mg/m2 IV bolus starting 1 hour into leucovorin infusion weekly for 6 weeks, repeated every 56 days).
- PG11047/Sunitinib: PG-11047 (infusion on Days 1 and 8 of a 21 day cycle) in combination with Sunitinib (50 mg orally once daily, 4 weeks on treatment followed by 2 weeks off (42 day cycle)).
Period: Overall Study
Arm/Group | PG11047/Gemcitabine | PG11047/Docetaxel | PG11047/Bevacizumab | PG11047/Erlotinib | PG11047/Cisplatin | PG11047/5-Flurouracil | PG11047/Sunitinib
Started | 12 | 9 | 34 | 34 | 48 | 32 | 3
Completed | 10 | 8 | 32 | 33 | 36 | 28 | 3
Not Completed | 2 | 1 | 2 | 1 | 12 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PG11047/Gemcitabine | PG11047/Docetaxel | PG11047/Bevacizumab | PG11047/Erlotinib | PG11047/Cisplatin | PG11047/5-Flurouracil | PG11047/Sunitinib | Total
Number analyzed (Participants) | 12 | 9 | 34 | 34 | 48 | 32 | 3 | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 26 | 20 | 31 | 20 | 1 | 110
  >=65 years | 4 | 5 | 8 | 14 | 17 | 12 | 2 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (10.8) | 63.2 (13.1) | 56.3 (12.8) | 62.8 (11.0) | 59.8 (10.1) | 60.2 (12.2) | 60.0 (24.4) | 59.8 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 15 | 18 | 19 | 14 | 2 | 80
  Male | 5 | 4 | 19 | 16 | 29 | 18 | 1 | 92
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 34 | 34 | 48 | 32 | 3 | 172

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the dose below which one-third of at least 6 patients (2/6) experienced a dose limiting toxicity (DLT).
  DLTs had to occur during cycle 1 of treatment and had to be considered related to PG-11047:
  1. Any nonhematologic toxicity > Grade 3 lasting > 3 days
  2. Grade 4 thrombocytopenia
  3. Grade 4 Anemia on the next scheduled dosing day
  4. Grade 4 Neutropenia (lasting > than 5 days
  5. Any febrile neutropenia (Grade 3 or 4))
  6. Inability to receive all scheduled doses of PG-11047 during the first dosing cycle due to drug related toxicity
Time Frame: End of Study
Population: Cohorts comprised 3 patients. When a patient experienced a treatment related toxicity qualifying as a DLT, up to 3 additional patients were to be enrolled at that dose. Patients who completed cycle 1 per protocol were evaluable.
Measure: Number; unit: mg
Groups:
- PG11047/Gemcitabine: PG-11047 in combination with Gemcitabine
- PG11047/Docetaxel: PG-11047 in combination with Docetaxel
- PG11047/Bevacizumab: PG-11047 in combination with Bevacizumab
- PG11047/Erlotinib: PG-11047 in combination with Erlotinib
- PG11047/Cisplatin: Cisplatin: 80 mg/m2 administered IV over 1 hour once every 28 days. PG-11047 will be administered on Days 1, 8 and 15 of a 28 day cycle.
- PG11047/5-Flurouracil: CGC-11047 in combination with 5-Flurouracil / Leucovorin
- PG11047/Sunitinib: PG-11047 in combination with Sunitinib.
  The MTD of PG-11047 was undetermineable due to only 2 evaluable patients in this treatment group
Arm/Group | PG11047/Gemcitabine | PG11047/Docetaxel | PG11047/Bevacizumab | PG11047/Erlotinib | PG11047/Cisplatin | PG11047/5-Flurouracil | PG11047/Sunitinib
Number analyzed (Participants) | 12 | 9 | 34 | 34 | 48 | 32 | 3
mg | NA — MTD not determined due to toxicities leading to study arm being prematurely stopped. | NA — MTD not determined due to toxicities leading to study arm being prematurely stopped. | 590 | 590 | 590 | 590 | NA — MTD not determined due to toxicities leading to study arm being prematurely stopped.

2. Secondary Outcome: Drug Safety
Time Frame: Ongoing
Reporting Status: Not Posted

3. Secondary Outcome: Pharmacokinetics
Time Frame: End of Study
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | PG11047/Gemcitabine | PG11047/Docetaxel | PG11047/Bevacizumab | PG11047/Erlotinib | PG11047/Cisplatin | PG11047/5-Flurouracil | PG11047/Sunitinib
Serious Adverse Events (participants affected / at risk) | 7/12 | 5/9 | 11/34 | 13/34 | 22/48 | 18/32 | 1/3
Other Adverse Events (participants affected / at risk) | 5/12 | 8/9 | 15/34 | 22/34 | 31/48 | 16/32 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PG11047/Gemcitabine (N=12) | PG11047/Docetaxel (N=9) | PG11047/Bevacizumab (N=34) | PG11047/Erlotinib (N=34) | PG11047/Cisplatin (N=48) | PG11047/5-Flurouracil (N=32) | PG11047/Sunitinib (N=3)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) — 2 not related and 1 unlikely related (Gemcitabine), 2 not related (Bevacizumab),1 related (cisplatin), 1 not related and 1 unlikely related (5-FU)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 4 (4) | 5 (5) | 0 (0) — Not related (2 Gemcitabine, 3 Bevacizumab, 2 Erlotinib, 4 Cisplatin, 5 5-FU)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 0 (0) — 2 unlikely related (Gemcitabine), 2 not related (Bevacizumab), 1 not related and 1 related (Erlotinib), 1 not related and 1 related (Cisplatin), 3 unlikely related (5-FU)
Altered mental status (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — 1 unlikely related (Gemcitabine), 1 not related (Erlotinib), 1 not related (Cisplatin)
Vomitting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0) — Not related (2 Gemcitabine, 1 Bevacizumab, 1 5-FU), unlikely related (1 Cisplatin, 2 5-FU), 2 related (Cisplatin)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — 1 not related (Gemcitabine) and 1 unlikely related (5-FU)
Uncontrolled pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Not related (Gemcitabine)
Right upper quadrant pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Not related (Gemcitabine)
Right lower chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Not related (Gemcitabine)
Bacteremia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — 1 not related (Gemcitabine), unlikely related (1 Gemcitabine, 1 5-FU)
Partial bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Not related (Gemcitabine)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — 1 not related and 1 related (Docetaxel)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) — Not related (1 Cisplatin, 1 Bevacizumab, 1 Erlotinib, 1 Cisplatin, 1 5-FU), unlikely related (1 Erlotinib)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (2) | 2 (2) | 0 (0) — Not related (3 Bevacizumab, 2 Cisplatin, 2 5-FU), unlikely related (1 Gemcitabine, 1 Erlotinib)
Neutroponic fever (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related (1 Docetaxel), related (1 5-FU)
Deep vain thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related (1 Docetaxel), related (1 Cisplatin)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — 1 not related and 1 unlikely related (Bevacizumab)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unlikely related (Bevacizumab)
Infection with normal ANC (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Not related (Bevacizumab)
Superventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related (1 Cisplatin), 1 unlikely related (Bevacizumab)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) — Not related (2 Erlotinib, 1 Cisplatin, 1 5-FU), related (1 Bevacizumab, 1 Cisplatin)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Not related (2 5-FU), unlikely related (2 Bevacizumab)
Pain right hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Not related (Bevacizumab)
Failure to thrive (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unlikely related (Bevacizumab)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5) | 2 (2) | 0 (0) — Not related (2 Erlotinib, 2 Cisplatin), unlikely related (1 Cisplatin, 2 5-FU), related (1 Erlotinib, 2 Cisplatin)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Unlikely related (Cisplatin)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unlikely related (Cisplatin)
Elevated creatinine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Related (Cisplatin)
Weakness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — 2 not related and 1 unlikely related (Cisplatin)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Not related (1 Cisplatin, 1 5-FU)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) — Not related (2 Cisplatin, 2 5-FU), unlikely related (1 Erlotinib)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Not related (1 Cisplatin), related (1 Erlotinib)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Not related (1 Cisplatin, 1 5-FU)
Oversedation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related (Cisplatin)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Not related and unlikely related (Cisplatin)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related (Cisplatin)
Unresponsive (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related (Cisplatin)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related (Cisplatin)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related (Cisplatin)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related (Cisplatin)
Elevated bilirubin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Not related (1 Erlotinib, 1 Cisplatin)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unlikely related (Cisplatin)
Pulmonary embolism (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) — Not related (2 Erlotinib, 1 Cisplatin), related (1 Cisplatin)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related (Cisplatin)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related (Cisplatin)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Unlikely related (1 Cisplatin), related (1 Cisplatin)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Not related (1 Cisplatin), unlikely related (1 5-FU)
Increased confusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Not related (1 Cisplatin, 1 5-FU)
Tracheostomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related (Cisplatin)
Post operative trachea hemorrhage (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related (Cisplatin)
Hypersensitivity allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related (Cisplatin)
Ureteral obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related (Cisplatin)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Not related (1 Cisplatin and 1 5-FU)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — Unlikely related (2 Cisplatin)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Not related (1 Erlotinib and 1Cisplatin)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related (Cisplatin)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Not related (1 Erlotinib, 1 Cisplatin, 1 5-FU)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) — Unlikely related (2 5-FU), related (5-FU)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unlikely related (5-FU)
GI bleed (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unlikely related (5-FU)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unlikely related (5-FU)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related (5-FU)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related (5-FU)
Intestinal ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unlikely related (5-FU)
Volume depletion (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) — Unlikely related (1 Erlotinib, 2 5-FU)
Ogilvie syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related (5-FU)
Acute CVA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related (5-FU)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related (5-FU)
Esophageal ulcers (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related (5-FU)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related (Erlotinib)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unlikely related (Erlotinib)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Related (2 Erlotinib)
Metastatic rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related (Erlotinib)
Hemorrhage CNS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Related (Sunitinib)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PG11047/Gemcitabine (N=12) | PG11047/Docetaxel (N=9) | PG11047/Bevacizumab (N=34) | PG11047/Erlotinib (N=34) | PG11047/Cisplatin (N=48) | PG11047/5-Flurouracil (N=32) | PG11047/Sunitinib (N=3)
Fatigue (General disorders) | 2 (2) | 3 (7) | 2 (2) | 4 (4) | 11 (18) | 8 (11) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (6) | 5 (16) | 0 (0) | 0 (0) | 3 (12) | 3 (7) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 6 (12) | 8 (9) | 4 (5) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 2 (2) | 3 (4) | 0 (0) | 9 (16) | 2 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (6) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 5 (7) | 12 (14) | 2 (2) | 0 (0)
Dyspnoea (Cardiac disorders) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central line infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 6 (7) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 0 (0) | 3 (5) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 4 (9) | 4 (4) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (12) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 6 (7) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Blood amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Cerebral haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No